CLINICAL TRIAL: NCT03730740
Title: Phase II Study of Lenalidomide Maintenance After Salvage Therapy in Patients With Relapsed and/or Refractory Non-Hodgkin T-cell Lymphoma
Brief Title: Phase II of Lenalidomide After Salvage Therapy in R/R Non-Hodgkin T-cell Lymphoma
Acronym: Lemon-T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, MD, Ph.D, Division of Hematology-Oncology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04-010
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Relapsed and/or Refractory Non-Hodgkin T-cell Lymphoma
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Administer the study drug in the following way with 28 days as one cycle. Lenalidomide 25mg Days 1-21 Dosing continues until disease progression is confirmed.
  Interventions: Drug: Lenalidomide 25mg

INTERVENTIONS:
Drug: Lenalidomide 25mg — Lenalidomide 25mg, day 1 - day 21 (1cycle=28days) for 2yeas
  Other Names: Lenalidomide

SUMMARY:
This study is to evaluate the efficacy and safety of lenalidomide maintenance therapy in patients with T-cell lymphoma who have undergone more than one treatment or relapsed after treatment and who acquired a response of more than a partial response after rescue chemotherapy. This is a phase 2 clinical trial.

DETAILED DESCRIPTION:
T-cell lymphoma that has relapsed after primary treatment or is refractory to treatment generally requires salvage therapy. In case of partial or complete response to such salvage therapy (partial response is determined by CT), consolidation therapy is performed to maintain the response and prevent relapse and autologous stem cell transplantation after high-dosage chemotherapy is generally adopted. However, autologous stem cell transplantation is unavailable if patient is over 65 years of age or not in a good full-body condition and additional treatment plans are required to prevent relapse in such cases. Allogenic stem cell transplantation after salvage therapy is also available in limited events in case of relapse after autologous stem cell transplantation and the effect of allogenic stem cell transplantation still not definite but experimental.

As a result, the treatment results of T-cell lymphoma that has relapsed are very poor despite active application of salvage therapy and overall survival (OS) and progression-free survival (PFS) have only been 5.5 and 3.1 months as a result of a previous study on 153 patients. Also, 3-year PFS after primary relapse was reportedly 16%. Likewise, overall survival (OS) of patients with T-cell lymphoma who experienced relapse or progression within first 24 months of diagnosis was 4.9 months (95% CI: 3.8-5.9 months). Therefore, additional therapy strategies are required to prevent relapse or progression of disease in patients who received salvage therapy for relapsed and/or refractory T-cell lymphoma.

Recently, the results of phase 2 study were reported where progressive survival period was effectively extended with Lenalidomide Maintenance for patients with relapsed and/or refractory diffuse large B cell lymphoma in cases where autologous stem cell transplantation is unattainable after salvage therapy.

Lenalidomide controls the immune system to activate the T cells or NK cells in the microenvironment of tumor for anti-tumor effects. Also, it combines with cerebron to lower IKZF1 and IKZF3 and inhibit MYC through the NF-kB route. MYC inhibition by Lenalidomide eventually lowers IRF4 to increase apoptosis and inhibit cell proliferation and induce anti-cancer effect accordingly . As a result, Lenalidomide was recognized as a treatment for multiple myeloma and lymphoma.

The results of clinical studies on the effect of Lenalidomide for T-cell lymphoma are still limited, but 26% OS has been reported for patients with T-cell lymphoma as a result of phase 2 clinical test where 25 mg (Day 1 - Day21, every 28 days) Lenalidomide was used as the only drug. Also, it has been proven that the increase of IRF4/MUM1, one of the major targets of Lenalidomide, is related to the poor prognosis of T-cell lymphoma, so the effect of Lenalidomide can be expected for T-cell lymphoma. Therefore, this study was conducted to evaluate the efficacies and safety of Lenalidomide Maintenance on patients who have shown partial response or complete response to salvage therapy for T-cell lymphoma that have been progressive after one or more therapies or relapsed after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The following subtypes of T-cell lymphoma histologically diagnosed based on WHO classification:

   * Peripheral T-cell lymphoma, not otherwise specified
   * Angioimmunoblastic T-cell lymphoma
   * Anaplastic large cell lymphoma, ALK-/+
   * Enteropathy-associated T-cell lymphoma
   * Monomorphic epitheliotropic intestinal T-cell lymphoma
   * Subcutaneous panniculitis-like T-cell lymphoma
   * Cutaneous T-cell lymphoma including mycosis fungoides and sezary syndrome
2. Relapse or progression after one or more previous therapies.
3. Partial response or more to a salvage therapy and at least 4 cycles of that salvage therapy at the time of participation in the clinical study.
4. Where autologous stem cell transplantation is unattainable due to poor physical conditions over 65 years of age or secondary transplantation is unattainable due to relapse after primary autologous stem cell transplantation.
5. Non-pregnant female patients who satisfy the following:

   - Natural menopause for at least 24 consecutive months before registering for the study or patients who had undergone hysterectomy or bilateral oophorectomy.
6. Male patients who can satisfy the following even if they are surgically infertile (with vasectomy):

   * Men must use an effective method of contraception during participation in the clinical test and for up to 4 weeks after administration.
   * Men must use condoms during administration of clinical drug, during temporary suspension of dosage, and for up to 4 weeks after administration if their partners are pregnant and not using an appropriate form of contraception (even after vasectomy).
   * Men must not donate their sperms during administration of clinical drug and for up to 4 weeks after administration and must immediately notify the researchers if their partners are pregnant during administration of clinical drug or right after suspending administration.
   * Must comply with the control plans for Lenalidomide (Appendix G).
7. 0 - 2 points in performance ability based on the classification of the eastern Cooperative Oncology Group (ECOG).
8. Appropriate condition of bone marrow, kidney, and liver.

   * White blood cells ≥ 4,000/μL
   * Neutrophes ≥ 1,500/μL
   * Platelets ≥ 75,000/μL (possible if ≥ 50,000/μL in case of intrusion in bone marrow)
   * Hemoglobin ≥ 9.0 g/dL (examination value is possible after correction through blood transfusion.)
   * Total bilirubin ≤ 1.5 x normal max.
   * AST/ALT ≤ 2.5 x normal max.
   * Creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula)
9. If the impact of all toxicity from the previous therapy is below Grade 1 based on Common Terminology Criteria for Adverse Events, Version 4.03.
10. Patients who are thought to perform and comply with the clinical test plan based on researcher's judgment.
11. Patients who have voluntarily agreed to participate in the clinical test and signed the consent.
12. Patients who have agreed to donate tissue slides and peripheral blood samples for participation in the clinical study.
13. In case of healthy Type B hepatitis carriers, patients are participatory if they can also undergo preventive antiviral treatment.

Exclusion Criteria:

1. Anyone classified into a histological subtype outside the selection criteria;
2. When autologous or allogenic stem cell transplantation is planned after salvage therapy;
3. Patients with symptomatic or uncontrolled angina pectoris or congestive heart failure, arrhythmia requiring chemotherapy, or major hazards anticipated due to clinically significant myocardial infarction that occurred 6 months in prior to participating in this clinical test;
4. In case of an infection exceeding Grade 2 under Common Terminology Criteria for Adverse Events, Version 4.03;
5. Anyone with an accompanied disease that is severe and uncontrolled;
6. Anyone with uncontrolled active Type B or C hepatitis (excluding healthy Type B hepatitis carriers who can be controlled by preventive antiviral agents);
7. Anyone infected with human immunodeficiency virus (HIV);
8. Anyone with allogenic organ transplantation or allogenic stem cell transplantation;
9. Anyone with history of a malignant tumor excluding the following diseases:

   * Anyone who has not received treatment for the target tumor or has not had any disease at least for the past 5 years; and
   * Anyone who has spent at least 1 year since complete removal of basal cell carcinoma/squamous cell carcinoma or successful treatment of cervical intraepithelial neoplasia;
10. Serious gastrointestinal bleeding exceeding Grade 2 under Common Terminology Criteria for Adverse Events, Version 4.03 within 30 days before screen;
11. Thrombosis or embolism within 6 months before screen;
12. If it is impossible to administer the clinical drug due to intrusion into the central nervous system (except for cases where the drug can be administered;
13. Any patient who is hypersensitive to this drug or a substance in this drug (ex: angioedema, Stevens-Johnson syndrome, toxic epidermal necrolysis, etc.);
14. Anyone with genetic problems, including galactose intolerance, Lapp lactase deficiency, and glucose-galactose malabsorption;
15. Anyone in an unstable state that may harm a patient's safety and compliance with the test;
16. Any patient with seizure disorder that requires drug administration;
17. Any drug abuse or medical, mental, or social disorder that may affect a patient's participation in clinical test or evaluation of clinical test results; and
18. Women who may be pregnant:

    * Anyone who has not undergone hysterectomy or bilateral oophorectomy and has not reached natural menopause for at least 24 consecutive months (not including no menstruation after anti-cancer treatment) (in that words, had menstruation anytime within the past 24 months).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Non-progressive survival period | 1 year
  The incidence of tumor progression or death from any cause up to 1 year from the first test drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Won-seog Kim, MD, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No